CLINICAL TRIAL: NCT05748561
Title: Effect of Intravenous Methylprednisolone and Intravenous Erythropoietin in Toxic Optic Neuropathies: Randomized Clinical Trial.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-22-02
Record Dates: First submitted 2023-02-20; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Toxic Optic Neuropathy; Treatment; Methylprednisolone; Erythropoietin
Keywords: Toxic Optic Neuropathy; Methylprednisolone; Erythropoietin
MeSH Terms: conditions — Toxic Optic Neuropathy | interventions — Methylprednisolone Hemisuccinate; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized groups (2)
  1. Standard treatment (Intravenous methylprednisolone)
  2. Intervention (Intravenous erythropoietin)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants won't be aware to which group they were assigned. Investigator in charge of assessing outcomes and analyzing data won't be aware to which group participants were assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patients will receive intravenous erythropoietin - 10,000 IU every 24 hours for 5 days.
  Interventions: Drug: Recombinant human erythropoietin 4,000 UI and 2,000 UI
- Control group (Placebo Comparator): The patients will receive intravenous methylprednisolone - 1 g every 24 hours for 5 days.
  Interventions: Drug: Methylprednisolone succinate 500 mg

INTERVENTIONS:
Drug: Recombinant human erythropoietin 4,000 UI and 2,000 UI — Intravenous recombinant human erythropoietin (10,000 IU every 24 hours for 5 days)
  Other Names: Experimental Group
  Arms: Experimental group
Drug: Methylprednisolone succinate 500 mg — Intravenous Methylprednisolone succinate (1 g daily for 5 days)
  Other Names: Control Group
  Arms: Control group

SUMMARY:
The goal of this double-blind prospective randomized clinical trial is to determine if the effect of intravenous erythropoietin is superior to the effect of intravenous methylprednisolone in cases of toxic optic neuropathy 4 weeks after therapeutic intervention.

The main question it aims to answer:

• Is there a difference in the visual recovery of toxic optic neuropathies treated with intravenous methylprednisolone in comparison with those treated with intravenous erythropoietin?

DETAILED DESCRIPTION:
A double-blind prospective randomized clinical trial of treatment for toxic optic neuropathies comparing visual outcome of patients treated by standard treatment (intravenous methylprednisolone) vs intravenous erythropoietin.

Enrollment: 18. Randomized groups (2)

1. Standard treatment (intravenous methylprednisolone)
2. Intravenous erythropoietin

Masking: Double (participant and outcomes assessor) Participants won't be aware to which group they were assigned. Investigator in charge of assessing outcomes and analyzing data won't be aware to which group participants were assigned

ELIGIBILITY:
Inclusion Criteria:

* Both genres.
* Age between 18 and 75 years.
* Clinical diagnosis of toxic optic neuropathy (afferent pupillary defect, acquired dyschromatopsia, visual loss and bilateral prechiasmatic field defect).
* Exposure with a temporal relationship of less than two weeks to a known toxicant for the function of the optic nerve.
* Up to 21 days from symptom onset.
* Informed consent signature.

Exclusion Criteria:

* History of previous optic neuropathy.
* History of additional ophthalmological or neurological pathology that has caused permanent visual loss.
* History of previous treatment with intravenous methylprednisolone or some other experimental treatment since the onset of symptoms.
* Poorly controlled diabetes mellitus.
* Poorly controlled systemic arterial hypertension.
* Hemoglobin >16 mg/dL
* Patients with a history of thromboembolic event.
* Patients with a history of coronary heart disease, myocardial infarction or cerebral vascular event.
* Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-04-05 (Estimated); Study Completion 2024-04-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Visual Capacity | Initial visit, 2-week visit, 1-month visit, 3-month visit
  Best corrected visual acuity

SECONDARY OUTCOMES:
Change from Baseline Color vision | Initial visit, 2-week visit, 1-month visit, 3-month visit
  Color vision as measured by Ishihara plates
Change from Baseline Visual field defect | Initial visit, 2-week visit, 1-month visit, 3-month visit
  Visual fields as measured by Goldmann perimetry
Change from Baseline Oct pRNFL (microns) | Initial visit, 3-month visit
  Nerve fiber thickness as measured by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cárdenas-Belaunzarán, MD, MSc, Study Director — Asociación Para Evitar la Ceguera en México I.A.P; Elsa Hernández-Piñamora, MD, Principal Investigator — Asociación Para Evitar la Ceguera en México I.A.P; Octavio Turcio-Aceves, MD, Principal Investigator — Asociación Para Evitar la Ceguera en México I.A.P
Locations (1):
- Jorge Cárdenas Belaunzarán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
This study is confidential and no information will be shared with the participants.

REFERENCES:
- [Background] Behbehani R. Clinical approach to optic neuropathies. Clin Ophthalmol. 2007 Sep;1(3):233-46. PMID 19668477
- [Background] Grzybowski A, Zulsdorff M, Wilhelm H, Tonagel F. Toxic optic neuropathies: an updated review. Acta Ophthalmol. 2015 Aug;93(5):402-410. doi: 10.1111/aos.12515. Epub 2014 Aug 27. PMID 25159832
- [Background] Karimi S, Arabi A, Shahraki T. Alcohol and the Eye. J Ophthalmic Vis Res. 2021 Apr 29;16(2):260-270. doi: 10.18502/jovr.v16i2.9089. eCollection 2021 Apr-Jun. PMID 34055263
- [Background] Kraut JA, Kurtz I. Toxic alcohol ingestions: clinical features, diagnosis, and management. Clin J Am Soc Nephrol. 2008 Jan;3(1):208-25. doi: 10.2215/CJN.03220807. Epub 2007 Nov 28. PMID 18045860
- [Background] Tan H, Kang X, Zhong Y, Shen X, Cheng Y, Jiao Q, Deng L. Erythropoietin upregulates growth associated protein-43 expression and promotes retinal ganglion cell axonal regeneration in vivo after optic nerve crush. Neural Regen Res. 2012 Feb 5;7(4):295-301. doi: 10.3969/j.issn.1673-5374.2012.04.010. PMID 25806072
- [Background] Sharpe JA, Hostovsky M, Bilbao JM, Rewcastle NB. Methanol optic neuropathy: a histopathological study. Neurology. 1982 Oct;32(10):1093-100. doi: 10.1212/wnl.32.10.1093. PMID 6889696
- [Background] Naeser P. Optic nerve involvement in a case of methanol poisoning. Br J Ophthalmol. 1988 Oct;72(10):778-81. doi: 10.1136/bjo.72.10.778. PMID 3191081
- [Background] Sun Y, Calvert JW, Zhang JH. Neonatal hypoxia/ischemia is associated with decreased inflammatory mediators after erythropoietin administration. Stroke. 2005 Aug;36(8):1672-8. doi: 10.1161/01.STR.0000173406.04891.8c. Epub 2005 Jul 21. PMID 16040592
- [Background] Pakdel F, Sanjari MS, Naderi A, Pirmarzdashti N, Haghighi A, Kashkouli MB. Erythropoietin in Treatment of Methanol Optic Neuropathy. J Neuroophthalmol. 2018 Jun;38(2):167-171. doi: 10.1097/WNO.0000000000000614. PMID 29300238
- [Background] Sharma R, Marasini S, Sharma AK, Shrestha JK, Nepal BP. Methanol poisoning: ocular and neurological manifestations. Optom Vis Sci. 2012 Feb;89(2):178-82. doi: 10.1097/OPX.0b013e31823ee128. PMID 22127151
- [Background] Pakravan M, Esfandiari H, Sanjari N, Ghahari E. Erythropoietin as an adjunctive treatment for methanol-induced toxic optic neuropathy. Am J Drug Alcohol Abuse. 2016 Nov;42(6):633-639. doi: 10.1080/00952990.2016.1198800. Epub 2016 Jul 27. PMID 27463192
- [Background] Kashkouli MB, Pakdel F, Sanjari MS, Haghighi A, Nojomi M, Homaee MH, Heirati A. Erythropoietin: a novel treatment for traumatic optic neuropathy-a pilot study. Graefes Arch Clin Exp Ophthalmol. 2011 May;249(5):731-6. doi: 10.1007/s00417-010-1534-3. Epub 2010 Oct 2. PMID 20890611
- [Background] Entezari M, Esmaeili M, Yaseri M. A pilot study of the effect of intravenous erythropoetin on improvement of visual function in patients with recent indirect traumatic optic neuropathy. Graefes Arch Clin Exp Ophthalmol. 2014 Aug;252(8):1309-13. doi: 10.1007/s00417-014-2691-6. Epub 2014 Jul 2. PMID 24986593
- [Background] Shayegannejad V, Shahzamani S, Dehghani A, Dast Borhan Z, Rahimi M, Mirmohammadsadeghi A. A double-blind, placebo-controlled trial of adding erythropoietin to intravenous methylprednisolone for the treatment of unilateral acute optic neuritis of unknown or demyelinative origin. Graefes Arch Clin Exp Ophthalmol. 2015 May;253(5):797-801. doi: 10.1007/s00417-014-2925-7. Epub 2015 Jan 22. PMID 25605544
- [Background] Feizi S, Alemzadeh-Ansari M, Karimian F, Esfandiari H. Use of erythropoietin in ophthalmology: a review. Surv Ophthalmol. 2022 Mar-Apr;67(2):427-439. doi: 10.1016/j.survophthal.2021.06.002. Epub 2021 Jun 23. PMID 34157346